CLINICAL TRIAL: NCT00306033
Title: IVIG Treatment Compared to Placebo in Patients With Myasthenia Gravis: A Randomized Clinical Trial
Brief Title: Intravenous Immune Globulin Treatment Compared to Placebo in Patients With Myasthenia Gravis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 03-0712-B
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Last update posted 2006-04-03 (Estimated); Status verified 2005-05

CONDITIONS: Myasthenia Gravis
Keywords: myasthenia gravis; immunoglobulin; intravenous immunoglobulin; treatment
MeSH Terms: conditions — Myasthenia Gravis

INTERVENTIONS:
Drug: Intravenous ImmuneGlobulin

SUMMARY:
This study is a double-blind, placebo-controlled, randomized clinical trial to determine whether IVIG is effective in improving motor scores in patients with myasthenia gravis and worsening weakness.

DETAILED DESCRIPTION:
Patients aged 18 years or older with a diagnosis of myasthenia gravis (MG) and worsening weakness were enrolled in the study after providing informed consent. Fifty-two patients were recruited to the study, but one withdrew consent prior to starting so that 51 patients were recruited. Baseline clinical assessments using the Quantitative MG Score for Disease Severity (QMGS) were repeated at 2 and 4 weeks after treatment with IVIG or saline infusion. The Post-Intervention Status was assessed at 2 and 4 weeks after treatment. The treatment was randomized and double-masked. Electrophysiological and immunological tests were done at baseline and after 2 weeks. Baseline characteristics were compared by the Student's t test for continuous variables or Chi-square test for categorical variables. An analysis of covariance was performed for the primary outcome measure, the change in QMGS.

ELIGIBILITY:
Inclusion Criteria:

* age > or equal to 18 years old with a confirmed diagnosis of myasthenia gravis and worsening weakness

Exclusion Criteria:

* age <18; severe myasthenia gravis requiring intensive care admission; change in immunosuppresive medication in previous 3 months; patients with severe bulbar weakness at risk for aspiration and respiratory failure; patients with other serious underlying medical conditions (renal failure, congestive heart failure); unwilling to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-03; Study Completion 2005-05

PRIMARY OUTCOMES:
change in the Myasthenia Gravis Foundation of America (MGFA) Quantitative MG Score for Disease Severity

SECONDARY OUTCOMES:
MGFA Post Intervention Status Scale, changes in single fiber eletromyography and repetitive nerve stimulation studies, changes in antiacetylcholine receptor antibody titers

CONTACTS AND LOCATIONS:
Overall Officials: Vera Bril, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada